CLINICAL TRIAL: NCT01813552
Title: A Phase I, Randomized, Open-label Study to Evaluate the Effect of Ritonavir or Omeprazole on the Pharmacokinetics of IDX719 in Healthy Subjects
Brief Title: To Evaluate the Effect of Ritonavir or Omeprazole on the Pharmacokinetics of Samatasvir (IDX719) in Healthy Participants (MK-1894-006)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1894-006; IDX-06A-006 (Other: Idenix Protocol Number)
Record Dates: First submitted 2013-03-13; First posted 2013-03-19 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Hepatitis C Infection
Keywords: HCV; Hepatitis C; antiviral drugs; liver
MeSH Terms: conditions — Hepatitis C | interventions — samatasvir; Omeprazole; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Samatasvir + Ritonavir (Experimental): Days 1, 9 and 13: Healthy Volunteers will take samatasvir in the mornings under fed or fasted conditions with water. Days 5-16: Healthy Volunteers will take ritonavir in the mornings under fasted or fed conditions with water.
  Interventions: Drug: Samatasvir; Drug: Ritonavir
- Samatasvir + Omeprazole (Experimental): Days 1, 9 and 13: Healthy Volunteers will take samatasvir in the mornings under fasted conditions with water or Coke. Days 5-16: Healthy Volunteers will take omeprazole in the mornings under fasted conditions with water or Coke.
  Interventions: Drug: Samatasvir; Drug: Omeprazole

INTERVENTIONS:
Drug: Samatasvir — Samatasvir 150 mg oral tablets (50mg x 3), single dose
Drug: Omeprazole — 40 mg delayed-release oral capsules, once daily
  Arms: Samatasvir + Omeprazole
Drug: Ritonavir — 100 mg oral tablets, once daily
  Arms: Samatasvir + Ritonavir

SUMMARY:
This study is designed to evaluate the potential for an effect of Ritonavir (Norvir®) or omeprazole (Prilosec®) on the pharmacokinetics of samatasvir and to assess the safety and tolerability of the study drugs when administered alone and in combination in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Read and signed the written informed consent form (ICF) after the nature of the study has been fully explained.
* All participants of childbearing potential must agree to use a double method of birth control (one of which must be a barrier) from Screening through at least 90 days after the last dose of the study drug.

Exclusion Criteria:

* Pregnant or breastfeeding.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter: Area under the concentration-time curve (AUC) from time zero to last measurable concentration | 0 hour (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, and 96 hours
Pharmacokinetic parameter: AUC from time zero to infinity | 0 hour (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, and 96 hours
Pharmacokinetic parameter: Maximum observed drug concentration (Cmax) | 0 hour (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, and 96 hours

SECONDARY OUTCOMES:
Percentage of participants who experienced at least one serious adverse event | Up to 17 days
Percentage of participants who experienced at least one adverse event | Up to 17 days
Percentage of participants who experienced at least one Grade 1 - 4 laboratory abnormality | Up to 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC